CLINICAL TRIAL: NCT02070783
Title: The Effects of ARA290 on the Cognitive and Neural Processing of Emotions in Healthy Volunteers
Brief Title: Cognitive and Neural Effects of ARA290
Acronym: CONEARA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Willem Van der Does, Professor of Psychology, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2010-024364-18
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Depression
Keywords: depression; cognition; emotion perception; information processing
MeSH Terms: conditions — Depression | interventions — cibinetide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARA290 (Experimental): 11-amino acid, linear peptide ARA290; intravenous injection with 2 mg ARA290 (single dosage).
  Interventions: Drug: ARA290
- Placebo (Placebo Comparator): saline (NaCl 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARA290
  Arms: ARA290
Drug: Placebo
  Arms: Placebo

SUMMARY:
Studies on the hormone Erythropoietin (EPO) have indicated that EPO may have antidepressant properties. However, EPO may cause serious side-effects with repeated administration (thrombosis), which limits its usefulness as an antidepressant. ARA290 is a peptide that does not have the effects of EPO on blood cells but may still have its effect on brain function. In an attempt to replicate previous findings with (a single dose of) EPO in healthy volunteers, we study the effects of ARA290 on the cognitive and neural processing of emotions in healthy volunteers. We hypothesize that a single dose of ARA290 will lead to a positive shift in information processing compared to placebo, 7 days post-administration.

DETAILED DESCRIPTION:
SUMMARY Rationale: Studies on the cognitive and neuronal effects of a single administration of Erythropoietin (EPO) in healthy volunteers and in depressed patients have suggested that EPO may have antidepressant effects. Due to its haematopoietic effects, EPO may cause serious side-effects with repeated administration, which limits its usefulness as an antidepressant. ARA290 is a peptide that does not have the haematopoietic effects of EPO but may still have its neurotrophic effects.

Objective: To study the effects of ARA290 on the cognitive and neural processing of emotions in healthy volunteers 7 days post-administration.

Study design: Randomized double-blind placebo-controlled experiment. Study population: Male and female healthy volunteers, n= 36; 18-35 yr old. Intervention: One group receives a single dose of 2 mg ARA290, the other group receives placebo.

Main study parameters/endpoints:

1. Behavioral study: Performance on an Emotional Test battery (ETB) which has been shown sensitive to antidepressant administration in healthy volunteers. The ETB includes a measure of facial expression recognition, emotional memory and attentional vigilance.
2. Neuroimaging study: Neural processing of emotions, in particular amygdala, hippocampal and VMPFC response to viewing facial stimuli expressing negative versus positive emotions.

Nature and extent of the burden and risks and benefits associated with participation:

Risks: No adverse events have been associated with the administration of a single dose of 70 -2000 μg ARA290 among 36 individuals, with the exception of one individual (with an undisclosed significant prior history of fainting) who fainted shortly after the intravenous dose administration of 700 μg ARA290 and recovered without medical intervention. Fourteen individuals have participated in a multiple dosing study with no serious adverse effects. Single doses of ARA290 in patients with renal impairment did not raise a safety signal.

Burden: Minimal. Emotional information processing test battery, burden comparable with playing computer games. fMRI measurement.

Benefits: Probably none. Possibly transient and small improvement of mood state. Financial compensation for participating.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking
* Age 18-35
* Right-handedness
* BMI 18 to 33 kg/m2

Exclusion Criteria:

* Major physical illness, such as diabetes, thyroid disease, epilepsy, stroke, multiple sclerosis, pituitary disease, or any other serious medical condition.
* Any current or past psychiatric disorder, including subclinical claustrophobia if severe enough to cause anxiety during scanning.
* Using medication likely to interfere with the study, including OTC (over the counter) medication (e.g., St John's Wort) and benzodiazepines.
* Pregnancy or breastfeeding
* Use of any nicotine products or soft drugs (hash, marihuana) in the three months prior to the study
* Any hard drug use (including XTC) (lifetime)
* Alcohol use of more than 14 units per week or more than 4 units on any day during the week prior to the study or during the study period.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
performance on information processing test battery, particularly emotion recognition | 1 week
  Performance on an Emotional Test battery (ETB) which has been shown sensitive to antidepressant administration in healthy volunteers. The ETB includes a measure of facial expression recognition, emotional memory and attentional vigilance.

SECONDARY OUTCOMES:
• Performance on a task of working memory | 1 week

OTHER OUTCOMES:
Neural response to angry faces | 1 week
  Neural processing of emotions, in particular amygdala, hippocampal and ventromedial prefrontal cortex (VMPFC) response to viewing facial stimuli expressing a negative or positive emotion.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Van der Does, PhD, Principal Investigator — Leiden University
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Background] Brines M, Cerami A. Erythropoietin-mediated tissue protection: reducing collateral damage from the primary injury response. J Intern Med. 2008 Nov;264(5):405-32. doi: 10.1111/j.1365-2796.2008.02024.x. PMID 19017170
- [Background] Miskowiak KW, Vinberg M, Harmer CJ, Ehrenreich H, Kessing LV. Erythropoietin: a candidate treatment for mood symptoms and memory dysfunction in depression. Psychopharmacology (Berl). 2012 Feb;219(3):687-98. doi: 10.1007/s00213-011-2511-1. Epub 2011 Sep 23. PMID 21947319
- [Derived] Cerit H, Veer IM, Dahan A, Niesters M, Harmer CJ, Miskowiak KW, Rombouts SA, Van der Does W. Testing the antidepressant properties of the peptide ARA290 in a human neuropsychological model of drug action. Eur Neuropsychopharmacol. 2015 Dec;25(12):2289-99. doi: 10.1016/j.euroneuro.2015.09.005. Epub 2015 Sep 18. PMID 26431906